CLINICAL TRIAL: NCT02644733
Title: Lecturer in Critical Care Nursing Department
Brief Title: Effect of Different Body Position on Intraabdominal Pressure in Mechanically Ventilated Patients
Acronym: Ghada
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Shalaby, lecturer in critical care nursing department, Assiut University
Other Study IDs: Ghada22
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Intraabdominal Hypertension
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — Urinary Catheters

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: head of bed elevation 30 degree — the intraabdominal pressure will be measured by nasogastric tube when the head of bed elevated to 30 degree
  Other Names: HOB30
Procedure: urinary catheter — the intraabdominal pressure will be measured by urinary catheter when the patient in supine position
  Other Names: flat position

SUMMARY:
Measuring intraabdominal pressure in the semi-recumbent position and supine position.

DETAILED DESCRIPTION:
Each set of measurements of intraabdominal pressure included intra bladder and intragastric pressure in the supine position followed by the semi-recumbent position at head of bed 30. All four measurements were taken over a period of 5 to 10 min or less to reduce the possibility of changes in intraabdominal pressure over time. Three sets of readings were taken at least 4 h apart over a 24-h period.

ELIGIBILITY:
Inclusion Criteria:

older than 18 years of age. to be sedated mechanically ventilated and to have both a nasogastric tube and indwelling urine catheter in place

Exclusion Criteria:

* recent oesophageal, gastric or bladder surgery; patients who were moribund and unlikely to survive 24 h; patients who were pregnant and patients who were unable to lay flat for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult mechanically ventilated patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
determine the effect of different body position on the intraabdominal pressure | up to 24 hour
  the intraabdominal pressure will be measured by urinary catheter and nasogastric tube when the patient in semi-recumbent position at 30 head of bed elevation)

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Sh Khalaf, Lecturer, Principal Investigator — Assuit university hospital
Locations (2):
- Egypt (2):
  - Assuit university hospital, Asyut, Assuit
  - Faculty of Nursing, Egypt, Assuit

IPD SHARING:
Plan to Share IPD: Yes
the patient's assessment sheet will be used to collect the data by the researcher

REFERENCES:
- [Background] Rooban N, Regli A, Davis WA, De Keulenaer BL. Comparing intra-abdominal pressures in different body positions via a urinary catheter and nasogastric tube: a pilot study. Ann Intensive Care. 2012 Jul 5;2 Suppl 1(Suppl 1):S11. doi: 10.1186/2110-5820-2-S1-S11. Epub 2012 Jul 5. PMID 22873412